CLINICAL TRIAL: NCT06403267
Title: A Multicentre, Prospective, Randomized, Open Label, Blinded-Endpoint, Placebo-controlled, Single-dose Trial to Determine the Efficacy and Safety of NoNO-42 in Participants With Acute Ischemic Stroke Selected for Thrombolysis With or Without Endovascular Thrombectomy (ACT-42 Trial)
Brief Title: NoNO-42 Trial in Acute Ischemic Stroke Patients Selected for Thrombolysis With or Without Endovascular Thrombectomy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NoNO Inc. (Industry)
Collaborators: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NoNO42-02 (ACT-42)
Record Dates: First submitted 2024-04-26; First posted 2024-05-07 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Acute Ischemic Stroke
Keywords: Thrombolysis, Endovascular thrombectomy; Reperfusion; Neuroprotection; Neuroprotectant
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, open label, blinded-endpoint (PROBE) controlled single-dose adaptive trial
Masking Description: Potential bias will be reduced by the following steps:
  * allocation concealment: via online central randomization
  * trial participants will remain blinded to dose and treatment allocation and will not be informed until after database lock.
  * blinded endpoint assessment, at Days 30 and 90 central blinded assessors will contact the participants for mRS and EQ-5D-5L assessments.
  Clinical site staff, including the Principal Investigator (PI), sub-investigators, clinic site staff, and the Sponsor will not be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- NoNO-42 (Active Comparator): Randomized participants will be given a single, 2.6 mg/kg 20-minute intravenous dose of NoNO-42 with a target start time of less than 10 minutes from randomization.
  Interventions: Drug: NoNO-42
- Control (No Intervention)

INTERVENTIONS:
Drug: NoNO-42 — a single dose sterile 20 ml vial containing lyophilized powder for reconstitution containing 300 mg of NoNO-42 active ingredient.
  Arms: NoNO-42

SUMMARY:
ACT-42 is a domain of the ACT-GLOBAL platform (NCT06352632).

This trial is a Phase 2b, multicenter, prospective, randomized, open label, blinded-endpoint (PROBE) controlled single-dose adaptive trial.

A total of up to 600 male and female participants aged ≥ 18 to ≤ 90 years harboring an acute ischemic stroke who are eligible for an intravenous thrombolytic with or without endovascular thrombectomy therapy will be enrolled within 4.5 hours of stroke onset/last known well.

DETAILED DESCRIPTION:
Because AIS is a medical emergency, the trial is designed to enable the administration of standard-of-care treatments in order to save the life of the person concerned, restore good health and alleviate suffering.

A total of up to 600 male and female participants aged ≥ 18 to ≤ 90 years harboring an acute ischemic stroke who are eligible for an intravenous thrombolytic with or without endovascular thrombectomy therapy will be enrolled within 4.5 hours of stroke onset/last known well. Randomization will be 1:1 drug/placebo. Randomization will be stratified by large vessel occlusion (LVO) (yes/no) and a minimization algorithm to minimize the contribution of imbalances in baseline factors (age, sex, baseline NIHSS score). The design is adaptive with prospective rules for adaptive enrichment, in which enrollment may be restricted to participants without an LVO. LVO is defined as an occlusion of the intracranial ICA, M1 or proximal M2.

Randomized participants will receive/received an intravenous thrombolytic and be allocated to:

* the investigational group, a single, 2.6 mg/kg (up to a maximum of 300 mg) 20-minute intravenous dose of NoNO-42, with a target start time of less than 10 minutes from randomization or
* the control group, no trial specific intervention.

Day 90: All participants will be followed for 90 days (or until death if prior to 90 days) for efficacy and 30 days for safety. The end of the trial is defined as the date that all participants have completed their Day 90 contact.

1-Year follow Up: participants who completed the trial to Day 90 may be followed at 1 year for long-term efficacy.

One database lock and corresponding report for the trial to Day 90 and a separate database lock and analysis for the 1-year follow up are planned.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed or suspected acute ischemic stroke (AIS) selected for intravenous thrombolysis.
2. Onset (last-known-well) time to randomization time within 4.5 hours.
3. Ages ≥ 18 to ≤ 90 years.
4. Disabling stroke defined as a baseline National Institutes of Health Stroke Score (NIHSS) >5.
5. Confirmed or suspected symptomatic anterior circulation intracranial occlusion. Tandem extracranial carotid and intracranial occlusions are permitted.
6. Pre-stroke independent functional status in activities of daily living as judged by the enrolling physician. Patient must be living without requiring nursing care.
7. Consent process completed as per national laws and regulation and the applicable ethics committee requirements.

Exclusion Criteria:

1. Large extent early ischemic changes/infarct in the ischemic territory on qualifying imaging.
2. Any intracranial hemorrhage on qualifying imaging.
3. Unlikely to initiate study drug administration before arterial puncture in those selected for EVT.
4. Known/suspected pregnancy and/or lactation.
5. Systolic blood pressure < 90 mmHg
6. Known prior receipt of NoNO-42 for any reason, including prior enrolment in this trial.

8) Severe comorbid illness with life expectancy less than 90 days, or likely to prevent completing 90-day follow-up.

9) Long term care facility resident or prisoner 10) Participation in another clinical trial outside of the ACT-GLOBAL platform investigating a drug or medical device or a neuro-interventional or surgical procedure that is not considered as standard care in the 30 days preceding trial enrolment.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Reducing global disability in participants with acute ischemic stroke (AIS) | 90 days from intervention
  The primary outcome is the mRS at Day 90. The primary analysis of the primary outcome will be a "shift" analysis, which is an ordinal analysis across the mRS scale. The primary estimand is odds-ratio for a better outcome on the mRS scale for NoNO-42 compared to control.

SECONDARY OUTCOMES:
Improving excellent functional outcome | 90 days from intervention
  Proportion of participants with a mRS of 0-1 at Day 90
Reducing worsening of stroke | 90 days from intervention
  Proportion of participants exhibiting a worsening of their index stroke during hospitalization.
  Worsening of stroke is defined as (A) progression of the index stroke or symptomatic intracranial, or symptomatic intracranial hemorrhagic within the first 7-days after randomization, supported and confirmed by medical imaging that is (a) life-threatening requiring intervention and/or (b) results in increased disability as gauged by a ≥ 4-point increase from lowest NIHSS during initial hospitalization or (B) results in death from the index stroke (i.e., index stroke is judged to be the principal cause of death) within the first 21-days after randomization.
Improving functional independence | 90 days from intervention
  Proportion of participants with a mRS of 0-2 at Day 90.
Reducing mortality rate | 90 days from intervention
  Proportion of participant mortality over the 90-day trial period
Improving health-related quality of life | 90 days from intervention
  Health-related quality of life, as measured by the EQ-5D-5L at Day 90

OTHER OUTCOMES:
1 year Follow-up | 1 year post intervention
  Whenever possible, participants will be followed up to 1 year post stroke to determine the efficacy of NoNO-42 at 1 year post stroke in:
  • Reducing global disability in participants with acute ischemic stroke (AIS).- - proportion of participants with a shift of one or more categories to reduced functional dependence analyzed across the whole distribution of outcomes on the mRS Scale
  The secondary objectives are to determine the efficacy of NoNO-42 at 1 year post stroke in:
  * Improving excellent functional outcome - Proportion of participants with a mRS of 0-1 at 1-year.
  * Improving functional independence - Proportion of participants with a mRS of 0-2 at 1-year
  * Reducing mortality rate - Proportion of participant mortality over 1-year
  * Improving health-related quality of life - Health-related quality of life, as measured by the EQ-5D-5L at 1-year
Safety Outcome | 30 and 90 days post intervention
  safety of a single 2.6 mg/kg dose of intravenous NoNO- 42 based on:
  * Serious adverse events (SAEs) to Day 30 and
  * 90-day mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Bijoy Menon, MBBS, MD, Study Chair — University of Calgary
Locations (9):
- Canada (9):
  - University of Calgary - Foothills Medical Centre, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - University of Manitoba, Winnipeg, Manitoba
  - Hamilton General Hospital, Hamilton, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Unity Health Toronto, St. Michael's Hospital, Toronto, Ontario
  - Royal University Hospital, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No